CLINICAL TRIAL: NCT01374841
Title: Nonmyeloablative Hematopoietic Stem Cell Transplantation (SCT) for High-Risk Hematologic Malignancies With Related, HLA-Haploidentical Donors: A Phase II Trial of Immunosuppression With Cyclophosphamide Administered Before and After SCT
Brief Title: Hematopoietic Cell Transplantation for Patients With Hematologic Malignancies Using Related, HLA-Haploidentical Donors
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IEO S513/110; 2009-018083-94 (EudraCT Number)
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Hematologic Neoplasms
Keywords: Hematopoietic Stem Cell Transplantation; High-Risk Hematologic Neoplasms; Haploidentical Donors; Cyclophosphamide
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Cyclophosphamide; Hematopoietic Stem Cell Transplantation; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Stem Cell Transplant+Cyclophosphamide (Experimental): patients with high-risk hematologic malignancies will receive hematopoietic stem cell transplantation from haploidentical donors after treatment with cyclophosphamide
  Interventions: Drug: Cyclophosphamide; Other: Hematopoietic Stem Cell Transplantation,

INTERVENTIONS:
Drug: Cyclophosphamide — 14.5 mg/kg, IV qd on day -6 and -5 and 50 mg/kg, IV on day +3 and +4
  Other Names: Endoxan
Other: Hematopoietic Stem Cell Transplantation, — Hematopoietic Stem Cell Transplantation,
  Other Names: Stem cell transplantation

SUMMARY:
The purpose of this study is to determine if engraftment can be achieved safely in patients with high-risk hematologic malignancies who undergo non-myeloablative transplant with peripheral stem cells from Human Leukocyte Antigen (HLA) haploidentical donors with pre and post-transplant cyclophosphamide as immunosuppression.

DETAILED DESCRIPTION:
It is important to extend the option of nonmyeloablative, hematopoietic stem cell transplantation (HSCT) for potential therapy of hematologic malignancies to patients who do not have an HLA-matched donor. Almost all patients would have a related donor identical for one HLA haplotype (haploidentical) and mismatched at HLA-A, B or DR of the unshared haplotype. Thus far, nonmyeloablative HSCT from HLA-mismatched donors has been associated with a high rate of graft failure and graft-versus-host disease (GVHD). In this protocol, we will use a combination of immunosuppressive agents including cyclophosphamide administered before and after HSCT to facilitate engraftment and to delete highly alloreactive T-cell clones presumably involved in GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≤70 years old
* Eligible diagnoses:
* CML in AP
* AML with high-risk cytogenetics [del(5q)/-5, del(7q)/-7, abnormal 3q, 9q, 11q, 20q, 21q, 17p, t(6:9), t(9;22), complex karyotypes (≥3 abnormalities)] in CR1
* AML ≥ CR2; patients should have <5% marrow blasts at the time of transplant
* High-risk ALL defined as:

CR1 with high-risk cytogenetics t(9;22), t(8;14), t(4;11), t(1;19) for adult patients >4 wk to achieve CR1

≥ CR2 Patients should have <5% marrow blasts at the time of transplant

* MDS (>int-1 per IPSS) after ≥ 1 prior cycle of induction chemotherapy; should have<5% marrow blasts at the time of transplant
* MM Stage II or III patients who have progressed after an initial response to chemotherapy or autologous HSCT or MM patients with refractory disease who may benefit from tandem autologous-nonmyeloablative allogeneic transplant
* CLL, NHL or HD who are ineligible for autologous HSCT or who have resistant/refractory disease and who may benefit from tandem autologous nonmyeloablative allogeneic transplant.
* Patients who have received a prior allogeneic HSCT and who have either rejected their grafts or who have become tolerant of their grafts with no active GvHD requiring immunosuppressive therapy could be enrolled

Exclusion Criteria:

* Patients with suitably matched related or unrelated donors
* Patients with conventional transplant options (a conventional transplant should be the priority for eligible patients ≤ 50 yr of age who have a related donor mismatched for a single HLA-A, -B or DRB1 antigen)
* CNS involvement with disease refractory to intrathecal chemotherapy
* Presence of active, serious infection (e.g., mucormycosis, uncontrolled aspergillosis, tuberculosis)
* Karnofsky Performance Status < 60% for adult patients (Appendix A)
* Patients with the following organ dysfunction:

  * Left ventricular ejection fraction <35%
  * DLCO <35% and/or receiving supplemental continuous oxygen
  * Liver abnormalities: fulminant liver failure, cirrhosis of the liver with evidence of portal hypertension, alcoholic hepatitis, esophageal varices, hepatic encephalopathy, uncorrectable hepatic synthetic dysfunction as evidenced by prolongation of the prothrombin time, ascites related to portal hypertension, bacterial or fungal liver abscess, biliary obstruction, chronic viral hepatitis with total serum bilirubin >3 mg/dL or symptomatic biliary disease.
* HIV-positive patients
* Women of childbearing potential who are pregnant (β-HCG+) or breast feeding
* Fertile men and women unwilling to use contraceptives during and for 12 months post transplant
* Life expectancy severely limited by diseases other than malignancy
* Patients on any other investigational drug at time of enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-08; Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Donor engraftment | Day +84
  percentage of donor engraftment after 84 from baseline

SECONDARY OUTCOMES:
Incidence and severity of graft versus host disease | up to 200 days after the baseline
  Incidence and severity of graft versus host disease after 200 days from the baseline
Non-relapse-related mortality | Incidence and severity of graft versus host disease after 200 days from the baseline
  incidence of non-relapse-related mortality after 200 days from the baseline

CONTACTS AND LOCATIONS:
Overall Officials: Rocco Pastano, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

REFERENCES:
- [Background] Luznik L, Jalla S, Engstrom LW, Iannone R, Fuchs EJ. Durable engraftment of major histocompatibility complex-incompatible cells after nonmyeloablative conditioning with fludarabine, low-dose total body irradiation, and posttransplantation cyclophosphamide. Blood. 2001 Dec 1;98(12):3456-64. doi: 10.1182/blood.v98.12.3456. PMID 11719388
- [Result] O'Donnell PV, Luznik L, Jones RJ, Vogelsang GB, Leffell MS, Phelps M, Rhubart P, Cowan K, Piantados S, Fuchs EJ. Nonmyeloablative bone marrow transplantation from partially HLA-mismatched related donors using posttransplantation cyclophosphamide. Biol Blood Marrow Transplant. 2002;8(7):377-86. doi: 10.1053/bbmt.2002.v8.pm12171484.